CLINICAL TRIAL: NCT05548244
Title: Multi-level Mechanisms of Behavioral Activation Therapy for Adolescent Depression
Brief Title: Mechanisms of Behavioral Activation (BA)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Wade Edward Craighead, PhD, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00078545; 1R01MH126985-01A1 (NIH)
Record Dates: First submitted 2022-09-15; First posted 2022-09-21 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Depression
Keywords: Behavioral Activation; fMRI
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MDD patients (Experimental): Participants will be seen for a maximum of 16 sessions over 16 weeks. Two extra sessions will be allowed during treatment.
  Interventions: Behavioral: Behavioral Activation Therapy; Behavioral: Baseline assessment procedures

INTERVENTIONS:
Behavioral: Behavioral Activation Therapy — Participants will be seen for a maximum of 16 sessions of therapy focused on increasing rewarding behaviors (16 individual therapy sessions of 1-hour, 2 of which include the BSIS component) over 16 weeks. BA intervention includes monthly booster sessions offered throughout 6-month follow up. If needed, two extra sessions will be allowed during treatment.
  Other Names: BA Therapy
Behavioral: Baseline assessment procedures — Completion of the K-SADS and CDRS-R to assess MDD, and the Wechsler Abbreviated Scale of Intelligence - 2nd Edition to assess IQ.

SUMMARY:
The investigators will be comparing brain (neural) activation of depressed adolescent patients before, during and after a course of Behavioral Activation (BA) therapy using functional magnetic resonance imaging (fMRI). In particular, the project seeks to determine whether BA targets different neural mechanisms for behavioral avoidance associated with low motivation as compared to threat avoidance. A group of healthy controls will also be scanned as a comparator group for behavioral and imaging measures.

DETAILED DESCRIPTION:
The primary aim of this study is to investigate the behavioral and neurobiological factors predicting response to Behavior Activation (BA), a psychosocial treatment for Major Depressive Disorder (MDD), in adolescents.

The recruitment age pool will be adolescents ages 15-17. The investigators plan to recruit 40 healthy controls and 96 treatment-seeking adolescents for an overall sample of ~136 participants, Individuals who reach the age of majority (18) during the study will be re-consented as adults and allowed to continue participating in the study.

A healthy control group will be included to assess stability in behavioral and neuroimaging measures over the course of participation in the study.

The fMRI scan schedule will include three task-based sessions (baseline, after session 7, and after endpoint) and two (sessions 3 & 9). "behavioral-scheduling-in-the-scanner" sessions Primary results will focus on symptom change within patients and their association to measures of low motivation and threat avoidance.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adolescents ages 15-17;
* current MDD diagnosis as determined by K-SADS-PL,
* CDRS-R raw score > 45 (T-score > 65) at baseline;
* estimated full scale IQ > 80 as determined by the WASI-II;
* able to receive outpatient care;
* willing to not partake in other psychosocial treatments;
* not taking psychotropic medications in the two weeks (four weeks for fluoxetine) prior to consent, with the exception of psychostimulant medication prescribed for the treatment of ADHD.
* Additionally, depressed patients must have access to required technology (e.g. smart phone, tablet, or desktop computer) to complete the EMA portion of the study.
* Healthy controls cannot not meet criteria for MDD and their CDRS-R raw score must be below 28; T-score < 52).

Exclusion Criteria:

* Current or past diagnosis of bipolar, schizophrenia, schizophreniform, schizoaffective disorders, or psychosis NOS;
* current diagnosis of developmental disorder, severe conduct disorder, life-threatening anorexia, OCD, or autism-spectrum disorders;
* taking psychotropic medications prior to entry;
* estimated IQ < 80; alcohol/drug dependence or abuse within the last 3 months;
* potential/confirmed neurological disorder or epilepsy;
* claustrophobia;
* presence of a medical condition that precludes fMRI;
* endorsement of imminent and serious suicidality;
* medical conditions that take precedence over the presence of MDD;
* pregnancy;
* substance use (excluding nicotine) within two weeks of the fMRI scan;
* left-handedness;
* nicotine use within 3 hours of the fMRI scan;
* history of traumatic brain injury or of being unconscious for more than 30 minutes;
* a stimulant regime for ADHD which has changed within 30 days of the fMRI scan.
* Non-compliance (i.e. <70% completion) or inability (i.e. lack of smartphone device) to complete the 3 assessment periods of EMA.

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 136 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Change in Diagnostic Interview Status (CDRS-R) total score from baseline | Baseline, week 16 post intervention
  Change from baseline on the Children's Depression Rating Scale-Revised (CDRS-R) total score. CDRS-R Total score measures the presence and severity of depression in children. The scale consists of 17 items scored on a 1-to-5- or 1-to-7-point scale. A rating of 1 indicates normal functioning and a higher number indicates a greater degree of depression. The total sum of scores range from 17 to 113. Following on prior studies of adolescent MDD, a diagnosis of MDD and a CDRS-R score of 45 or greater is the criterion for admission to the study. A score of 27 or less at the end of the study is the criterion for remission of MDD.
Change in Adolescent Longitudinal Interval Follow-Up Evaluation (A-LIFE) | Week 8 post intervention (Midpoint), week 16 post intervention
  The A-LIFE Interview, developed for use with adolescents, was based on the Longitudinal Interval Follow-up Evaluation scale (LIFE), a clinical interview for adults. The A-LIFE comprises three general sections, including psychopathology, psychosocial functioning, and general severity of the disorder (GSD). The psychopathology domain will be used in the current study because it provides information regarding whether the participant has met the criteria and symptoms of DSM-5 disorders. The A-LIFE measure of greatest interest in the current study is the 6-point rating of each identified psychiatric disorder. Each form of psychopathology is scored 1-6, and a depression score of 4, 5, or 6 yields a positive diagnosis of MDD. The primary outcome variable will be the number of MDD patients reaching remission status (<4).

SECONDARY OUTCOMES:
Change in Beck Depression Inventory (BDI-II) | Baseline, weekly therapy visits 1-16 post intervention
  BDI-II is a 21-self report assessment of the level of depressive symptoms over 2-week period. The minimum and maximum values for the BDI-II are (0-63). The higher the scores, the greater the severity of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Wade E Craighead, PhD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory University, Atlanta, Georgia
  - Facility for Education and Research in Neuroscience (FERN), Atlanta, Georgia
  - Child and Adolescent Mood Program (CAMP), Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
De-identified data (including access and additional documents) will be shared through the NIMH NDA and in accordance with NIMH NDA data-sharing policy.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: As soon as possible after data collection.
Access Criteria: In accordance with NIMH NDA data-sharing policy.